CLINICAL TRIAL: NCT05715424
Title: Research on Precise Myopia Prevention and Control Technology and Demonstration Application for Children and Adolescent
Brief Title: Community Intervention and Demonstration Area Construction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: Shanghai Eye Disease Prevention and Treatment Center (Other); Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Fangbiao Tao, Professor and Dean, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20210735
Record Dates: First submitted 2022-11-10; First posted 2023-02-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Myopia; Refractive Errors
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cluster A (Experimental): The study population (school-based) was divided into four clusters.Each cluster will receive the same intervention.and one cluster was randomly selected as Cluster A. The intervention was administered at month 6 and monitored for two years.
  Interventions: Other: Six interventions for children and adolescents
- Cluster B (Experimental): The study population (school-based) was divided into four clusters. Each cluster will receive the same intervention.and one cluster was randomly selected as Cluster B. The intervention was administered at month 12 and monitored for one and a half years.
  Interventions: Other: Six interventions for children and adolescents
- Cluster C (Experimental): The study population (school-based) was divided into four clusters.Each cluster will receive the same intervention. and one cluster was randomly selected as Cluster C. The intervention was administered at month 18 and monitored for a continuous period of one year.
  Interventions: Other: Six interventions for children and adolescents
- Cluster D (Experimental): The study population (school-based) was divided into four clusters.Each cluster will receive the same intervention.and one cluster was randomly selected as Cluster D. The intervention was implemented at month 18 and an evaluation of the effect of the intervention was performed.
  Interventions: Other: Six interventions for children and adolescents

INTERVENTIONS:
Other: Six interventions for children and adolescents — * Vision Health Record Establishment and Myopia Risk Assessment.
  * Evaluation of vision care behavior and development of reasonable eye use behavior.
  * Health education for teachers and parents.
  * Action to improve the reading and writing environment at home and school.
  * One hour of outdoor activities in and out of school during the day.
  * Myopia grading management and medical correction action.

SUMMARY:
The objective of this intervention study was to understand the visual health status of nearly one million children and adolescents in ten provinces in China, and then to conduct intervention and evaluate the effect of intervention measures with the development of myopia as the outcome indicator. The study will be conducted in the form of a stepped intervention and will answer the following questions.

Current China children and adolescent's vision health, including the different degrees of myopia prevalence, and farsightedness reserve status. To evaluate the implementation and effect of eight appropriate technologies and six interventions developed in this study, to reduce the incidence of myopia among children and adolescents in China, to achieve the purpose of nationwide application.

In the early stage of this study, a baseline survey will be conducted on participants. In the middle stage, participants will be required to adjust the seat height regularly and increase the time for outdoor activities, etc. In the later stage, intervention measures will be evaluated based on the overall research situation to consider national promotion.

ELIGIBILITY:
Inclusion Criteria:

* ● Kindergarten kids.

  * Grade of 1 to 6 in elementary schools.
  * Grade of 1 to 3 in middle schools.
  * Grade of 1 to 3 in high schools.
  * Sign the informed consent.

Exclusion Criteria:

* ●Visual defect or other eye diseases.

  * wearing orthokeratology; refractive surgery history.
  * Not considered suitable for inclusion in the study by the investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in questionnaire survey | Baseline, 6 months, 1 year, 1.5 years, 2 years
  Questionnaires based on myopia prevention and control for children and adolescents, including a questionnaire on myopia in children and adolescents.
Changes in uncorrected vision within two years | Baseline, 6 months, 1 year, 1.5 years, 2 years
  Uncorrected visual acuity (UCVA) was measured for the right eye, then the left eye, with a E Standard Logarithm Vision Acuity Chart (GB11533-2011) in 5-grade notation (5- LogMAR), with illumination of the chart around 500lx. If one of the eyes UCVA was less than 5.0, then tests with combined lenses were conducted among the poor eye-sighted for confirming the types of ametropia (normal, myopia, hyperopia or other eye diseases)．All the measurements were recorded.
Changes in visual acuity in computer optometry | Baseline, 6 months, 1 year, 1.5 years, 2 years
  Optometry Automated computerized optometry is performed by an optometrist. Automatic optometry instrument using desktop computer automatic optometry, equipment requirements should conform to the "ISO10342-2010 Ophthalmic instruments: Optometry" provisions.
Changes in visual acuity during dilated pupil optometry | Baseline, 6 months, 1 year, 1.5 years, 2 years
  Between 5% and 10% of the participants were selected for Dilated pupil optometry.

SECONDARY OUTCOMES:
Eye protection diary | Three months.
  Daily questionnaire based on the development of myopia prevention and control in children and adolescents.
Qualitative interview | Baseline, 1 year, 2 years
  Based on the interview outline on myopia prevention and control, some randomly selected students, parents, teachers and related departments were investigated.

CONTACTS AND LOCATIONS:
Overall Officials: FangBiao Tao, Professor, Study Director — Anhui Medical University
Locations (1):
- Anqing myopia scene, Anqing, Anhui, China

IPD SHARING:
Plan to Share IPD: No